CLINICAL TRIAL: NCT03155126
Title: The Effect of Different Crystalloids on the Incidence of Acute Kidney Injury in Shock Patients
Brief Title: Different Crystalloids on AKI in Shock
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Attending Doctor, Southeast University, China
Other Study IDs: 2017ZDSYLL017P01
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Shock
Keywords: shock; acute kidney injury; crystalloid
MeSH Terms: conditions — Shock; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Saline group: Patients resuscitated with saline
  Interventions: Other: Fluid resuscitation
- Acetated Ringer's sodium group: Patients resuscitated with Acetated Ringer's sodium
  Interventions: Other: Fluid resuscitation

INTERVENTIONS:
Other: Fluid resuscitation — Patients in the saline group were resuscitated with saline, patients in the other group were resuscitated with acetated Ringer's sodium

SUMMARY:
The goal is to observe that the incidence of acute kidney injury in patients who need fluid resuscitation when resuscitated with saline or acetated Ringer's sodium.

DETAILED DESCRIPTION:
Fluid resuscitation is important to shock patients. Saline is the classical fluids for resuscitation. However, studies showed that resuscitation with saline could increase the incidence of hyperchloremia and acute kidney injury. Thus, the goal is to observe that the incidence of acute kidney injury in patients who need fluid resuscitation when resuscitated with saline or acetated Ringer's sodium.

ELIGIBILITY:
Inclusion Criteria:

* Shock patients who need fluid resuscitation with risk factors of acute kidney injury

Exclusion Criteria:

* Patients with a history of chronic kidney injury and hemodialysis therapy

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Shock patients who need fluid resuscitation with risk factors of acute kidney injury
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | 28 day
  Incidence of acute kidney injury

SECONDARY OUTCOMES:
Application of renal replacement | 28 day
  Application of renal replacement

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided